CLINICAL TRIAL: NCT02999724
Title: Gabapentin Reduces Opioid Use Postoperatively ("GROUP Study"): A Randomized Control Trial in Women Undergoing Reconstructive Pelvic Surgery
Brief Title: Gabapentin Reduces Opioid Use Postoperatively ("GROUP Study")
Acronym: GROUP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Danny Lovatsis, Dr., Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16-0262-A
Record Dates: First submitted 2016-12-17; First posted 2016-12-21 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- gabapentin (Experimental): gabapentin 300-600 mg 1 hour preop
  Interventions: Drug: Gabapentin
- placebo (Placebo Comparator): placebo capsule(s) 1 hour preop
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Gabapentin — Gabapentin 300-600 mg 1 hour preop
  Arms: gabapentin
Other: placebo — placebo capsule(s) 1 hour preop
  Other Names: placebo capsule
  Arms: placebo

SUMMARY:
Gabapentin is a medication used primarily to treat seizures and pain. Studies have shown that this medication can help reduce pain after surgery, including hysterectomy, where the uterus or "womb" is removed. Opioids are the first choice for pain medication administered after surgery, but carry significant side effects. Several studies have demonstrated that if patients are given gabapentin before surgery, they require less opioids after surgery. However, there have not been any studies examining gabapentin's effects on post-operative pain in urogynecologic surgery, which treats pelvic organ prolapse and urinary incontinence. Pelvic organ prolapse occurs when female pelvic floor supports have weakened and therefore patients experience a "bulge" or "pressure" in the vagina. Patients with these conditions are typically offered medical treatments, but some may require surgery, and this usually consists of vaginal hysterectomy, pelvic floor repair, and a mid-urethral sling to treat any concurrent urinary incontinence. Our study aims to look at the effect of gabapentin given to patients undergoing urogynecologic surgery on their pain levels after surgery, including the amount of opioid pain medication required. We hypothesize that the patients who receive gabapentin before surgery will require significantly less opioids.

Over a six-month period, patients seen in Urogynecology clinics will be invited to participate in the study. Women who are already on gabapentin for other reasons, have an allergy to gabapentin, have a reason they cannot take gabapentin, or who cannot understand spoken English will be excluded from the study. After providing informed consent, they will be randomized to either receive gabapentin or a placebo pill. They will receive the standard surgical care, including the usual anesthesia for surgery and routine pain medications available after surgery. We will then compare the differences in opioid consumption in the first 24 hours after surgery as well as the time from the end of surgery to leaving to the recovery room and the length of recovery room stay between the gabapentin and placebo groups. We will also analyze the differences in anxiety, drowsiness, pain, and nausea as rated by the patients in each group.

DETAILED DESCRIPTION:
This study will be a randomized double blinded placebo controlled trial. All women presenting to Mount Sinai Hospital eligible for surgery with pelvic organ prolapse symptoms requiring hysterectomy with other pelvic reconstruction (repair of cystocele and/or rectocele, with or without TVT) will be provided with a written informed consent to be randomized to either receiving pre-operative gabapentin single dose or placebo 2 hours prior to surgery. The single dose of gabapentin will be 600 mg for patients under 65 years old and 300 mg for those 65 years old and above. All patients will have pre-operative assessment according to the usual routine that will include urogynecological history taking, physical examination, urodynamic testing and blood work. Urodynamic testing will include measurement of the post-void residual by urethral catheterization or bladder scan, uroflowmetry, a filling cystometrogram and urethral pressure profilometry. Medication and placebo will be prepared by the hospital pharmacy to look alike to blind staff and patients. Medication or placebo will be given with other pre-anesthesia medications such as celecoxib and acetaminophen according to usual protocol. Routine peri-operative surgical/anesthesia management will be unchanged from the usual care. Post-operative pain score will be measured using a visual analogue scale (VAS) from 1 to 10. Total Opioids use during the first 24 hours after surgery will be calculated from patients' paper and electronic chart, and conversion will be made to morphine equivalents.

ELIGIBILITY:
Inclusion Criteria:

* women age 18 years and older
* uterovaginal prolapse with or without stress urinary incontinence
* booked for vaginal hysterectomy, anterior and/or posterior vaginal repair, with or without TVT

Exclusion Criteria:

* Women already on gabapentin for other indications
* Women with proven allergy or sensitivity to gabapentin
* Women with a contraindication to gabapentin
* Women unable to understand spoken English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-09 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
opioid consumption postop | 24 hours
  total opioid use 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Danny Lovatsis, MD, Principal Investigator — Sinai Health System
Locations (1):
- Department of Obstetrics and Gynecology, Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li ALK, Wadsworth K, Siddiqui NT, Alarab M, McDermott CD, Lemos N, Dawood A, Lovatsis D. Does low-dose gapapentin reduce opioid use postoperatively?: A randomized controlled trial in women undergoing reconstructive pelvic surgery. Int Urogynecol J. 2019 Feb;30(2):211-217. doi: 10.1007/s00192-018-3617-3. Epub 2018 Mar 21. PMID 29564507